CLINICAL TRIAL: NCT05941559
Title: Effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) Therapy in Rheumatoid Arthritis (RA) Patients With Persistent Pain Despite Inflammation Being Under Control: a Multiple Baseline Single Case Experimental Design Study Across Ten Cases
Brief Title: EMDR for Persistent Pain in RA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: University of Twente (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Harald E. Vonkeman, prof.dr., Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMDR in RA
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Chronic pain; EMDR
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Pain | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: A multiple-baseline single-case experimental design (SCED) across three time series. Participants will be randomized to one of the three time series. Within the time series the start of the intervention is randomly determined. Four participants will be assigned to the shortest, three to the medium and three to the longest baseline length. The SCED study consists of a baseline phase (A1), intervention phase (B), post-treatment phase (A2), follow-up phase 1 (A3), and follow-up phase 2 (A4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shortest baseline length (Other): Intervention starting points are at day 15, 16, 17, 18 or 19.
  Interventions: Other: EMDR
- Medium baseline length (Other): Intervention starting points are at day 20, 21, 22, 23, and 24.
  Interventions: Other: EMDR
- Longest baseline length (Other): Intervention starting points are at day 25, 26, 27, 28, or 29.
  Interventions: Other: EMDR

INTERVENTIONS:
Other: EMDR — Eye Movement Desensitization and Reprocessing

SUMMARY:
Rationale: Around 20% of rheumatoid arthritis (RA) patients have persistent pain, despite having well-controlled disease activity. There is a significant overlap in underlying mechanisms between post-traumatic stress disorder (PTSD) and persistent pain. Eye Movement Desensitization and Reprocessing (EMDR) is a proven effective treatment for PTSD and evidence is growing that it may also be effective for persistent pain. Objective: To assess the feasibility and estimate the effectiveness of EMDR in RA patients with persistent pain despite inflammation being under control.

Study design: A multiple-baseline single-case experimental design (SCED) across three time series. Participants will be randomized to one of the three time series. Within the time series the start of the intervention is randomly determined. Four participants will be assigned to the shortest, three to the medium and three to the longest baseline length. The SCED study consists of a baseline phase (A1), intervention phase (B), post-treatment phase (A2), follow-up phase 1 (A3), and follow-up phase 2 (A4).

Study population: Subjects are RA patients > 18 years with low disease activity (DAS28<3.2) at >2 measurements over the previous 12 months and concurrent elevated pain scores (NRS-pain>6).

Intervention (if applicable): EMDR therapy consists of an intake and eight sessions of 90 minutes in total, performed according to the EMDR standard protocol, conducted by four psychologists, all are level-II trained, under the supervision of an EMDR Europe consultant. EMDR focuses on processing traumatic memories, pain-related memories, and current physical pain.

Main study parameters/endpoints: Primary endpoint for effectiveness is the pre-treatment phase A1 to post-treatment phase A2 difference in NRS pain intensity. Feasibility is examined by monitoring recruitment, dropout rates, and treatment satisfaction. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: If the therapy is effective, pain intensity decreases, additional physical complaints of RA decrease and participants experience less discomfort from their pain in daily life. EMDR therapy is an evidence-based treatment for PTSD and the reduction of posttraumatic stress favors the recovery of physical complaints. Participating in the study includes two conversations for inclusion (two times 60 minutes consisting of one telephone conversation and one face-to-face conversation), attending the EMDR therapy intake (one time 90 minutes) and sessions (eight times 90 minutes), and daily registration of complaints (about two minutes per day) via a smartphone application, completing the questionnaires (about 14-28 minutes at six specific time points during the study), and an exit conversation at six months follow up. Daily registration will take 18 to 20 weeks maximum. At the three- and six-month follow-up, participants will be asked to register daily for 14 days. EMDR sessions can be emotionally intense, but never are as challenging as living with unprocessed (traumatic) pain-related memories. There are no risks associated with EMDR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RA
* Stable low disease activity Score in 28 joints, i.e. DAS28 <3.2 at >2 measurements over the previous 12 months and at the time of inclusion
* Elevated pain scores (NRS pain >6) at >2 measurements over the previous 12 months and at the time of inclusion
* Sufficient knowledge of the Dutch language

Exclusion Criteria:

* An acute condition of psychosis or bipolar disorder
* An acute suicidal risk
* Substance dependency
* Not stable on the use of medication
* Visual or hearing problems interfering with the EMDR procedure
* Other psychological/psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 100 Days
  Difference in Numeric Rating Scale (NRS) pain intensity. Scale 0-6, 0 means never (good outcome), 6 means always (bad outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided